CLINICAL TRIAL: NCT06771284
Title: Problem Behavior Assessment and Intervention in IDEA Part C Services: A Single-Case Study
Brief Title: Problem Behavior Assessment and Intervention in IDEA Part C Services
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Collaborators: Institute of Education Sciences (U.S. Federal Agency)
Responsible Party: Principal Investigator, Stephanie Gerow, Associate Professor, University of Nevada, Las Vegas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UNLV-2024-418
Record Dates: First submitted 2024-06-24; First posted 2025-01-13 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Problem Behavior; Developmental Delay; Developmental Disability
Keywords: Early childhood; Problem behavior; Home-based services; IDEA Part C services
MeSH Terms: conditions — Problem Behavior; Learning Disabilities; Developmental Disabilities | interventions — Methods

STUDY DESIGN:
Intervention Model Description: The investigators will use a multiple baseline design across participants with a baseline and intervention phase to evaluate the effects of the intervention on children's challenging behavior. Each of the 3 tiers of the multiple baseline will include a caregiver-child dyad. One early intervention professional will work with each caregiver-child dyad, for a total of 9 participants across 3 tiers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Following baseline (i.e., no intervention/business as usual) sessions, children will receive the intervention, consisting of a function-based intervention. This intervention will be implemented by the caregiver. The intervention will consist of teaching the child an alternative, appropriate skill (usually communication) to replace the problem behavior. The caregiver will provide reinforcement for the appropriate skill and no reinforcement (i.e., extinction) following problem behavior. The caregiver will also learn and use general strategies for teaching social-emotional skills (e.g., setting appropriate rules) as part of the intervention.
  Interventions: Behavioral: Function-based assessment and intervention

INTERVENTIONS:
Behavioral: Function-based assessment and intervention — This intervention will be implemented by the caregiver. The intervention will consist of teaching the child an alternative, appropriate skill (usually communication) to replace the problem behavior. The caregiver will provide reinforcement for the appropriate skill and no reinforcement (i.e., extinction) following problem behavior. The caregiver will also learn and use general strategies for teaching social-emotional skills (e.g., setting appropriate rules) as part of the intervention.

SUMMARY:
The purpose of this study is to evaluate the effect of function-based assessment and intervention to reduce problem behavior in children with developmental disability or delay in the context of IDEA Part C services. The investigators will conduct a single-case study to evaluate the efficacy of the intervention.

ELIGIBILITY:
Child Inclusion Criteria:

* age birth to 5 years old
* has a developmental disability or delay based on caregiver report and/or receiving early intervention services
* has problem behavior, as reported by the caregiver and/or early intervention professional

Caregivers (e.g., parent, grandparent) of eligible child participants will participate with their child as the implementer of all procedures.

An early intervention professional will participate with each caregiver-child dyad to coach the caregiver, in addition to the researcher.

Ages: 0 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 9 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Problem Behavior | The investigators plan to conduct approximately weekly observations, with a total of 15 observations.
  The investigators will conduct 5-min observations and record the frequency of the child's problem behavior (e.g., aggression, self-injury, screaming) during each session. The specific problem behavior(s) recorded will be defined individually by participant.

SECONDARY OUTCOMES:
Appropriate Behavior | The investigators plan to conduct approximately weekly observations, with a total of 15 observations.
  The investigators will conduct 5-min observations and record the frequency of the child's appropriate behavior (e.g., communication) during each session. The specific appropriate behavior(s) recorded will be defined individually by child participant.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nevada Las Vegas, Las Vegas, Nevada, United States